CLINICAL TRIAL: NCT03258073
Title: Impact of Simulation Scenario Execution on Acute Care Skills and Confidence Related to Maternal and Pediatric Care Emergencies Among Pre-service Health Professional Trainees in Uganda
Brief Title: Does Simulation Scenario Execution Improve Acute Care Skills and Confidence Related to Maternal and Pediatric Care Emergencies?
Acronym: SimForLife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MUST 21/06-16b
Record Dates: First submitted 2017-08-14; First posted 2017-08-23 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Maternal, Pediatric Care Emergencies
Keywords: maternal; newborn; resuscitation; emergencies; medical simulation
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Investigators will conduct a cohort study among medical and nursing students and follow groups of students according to their rotation in the four major clinical disciplines. A cohort will represent a group of students who start a clinical rotation and complete their clinical year together. A total of 4 rotations exist concurrently every academic year in a year of study (Pediatrics, Internal medicine, Surgery and Obstetrics). During each rotation, a cohort will be exposed to at least 1 simulation scenario relevant to the discipline of the rotation. Investigators hypothesize that repeated exposure to simulation scenario execution will improve CTS scores. Therefore in this cohort study, investigators will measure CTS scores before and after exposure to simulation scenario training.
Masking Description: No masking will be done
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical simulation using scenarion execution (Experimental): Study participants will be exposed to medical simulation using scenario execution. In this exercise, participants will be exposed to a scenario that simulates a medical emergency. They will be required to respond. Following their response, the participants will have a chance to share with the investigators their experiences and what they have learnt from the exposure in a debriefing session. The investigator will then provide feedback on their performance.
  Interventions: Other: Medical simulation using scenario execution

INTERVENTIONS:
Other: Medical simulation using scenario execution — Each team of students will be exposed to simulation two times in a semester totaling to four times a year. In a scenario execution, participants are placed in a simulated experience of a medical emergency. Participants are required to respond and their reactions are observed by the investigators. After the experience, participants will have a debriefing session to learn from their experience of handling this emergency.
  Other Names: medical simulation methodology

SUMMARY:
In Uganda and many countries in Sub-Saharan Africa, health providers have minimal training and intermittent opportunity to maintain skills in managing delivery complications and acute newborn and pediatric conditions. Interventions like effective resuscitation assistance at the time of birth are lifesaving. Every 30 second delay in establishing effective resuscitation at birth increases the risk of death by 16%. The purpose of this study is to test whether medical simulation can improve acute care skills and confidence related to maternal and pediatric care emergencies.

DETAILED DESCRIPTION:
In Uganda and many countries in Sub-Saharan Africa, health providers have minimal training and intermittent opportunity to maintain skills in managing delivery complications and acute newborn and pediatric conditions. Interventions like effective resuscitation assistance at the time of birth are lifesaving. Every 30 second delay in establishing effective resuscitation at birth increases the risk of death by 16%. The purpose of this study is to test whether medical simulation can improve acute care skills and confidence related to maternal and pediatric care emergencies.

A solid body of evidence now supports simulation-based learning as superior to didactic teaching and problem-based learning for the acquisition of critical assessment and management skills, particularly for clinical emergencies. Simulation-based training promotes skill acquisition and retention, enhances teamwork, and increases knowledge and understanding of key procedures. Simulation-based learning is now the norm in medical, nursing and paramedical training in most high income settings. There remains a critical need to operationalize simulation-based learning in resource-constrained settings

ELIGIBILITY:
Inclusion Criteria:

* Participants are medical and nursing students in active clinical rotation; third and fifth year medical students and third and fourth year nursing students at Mbarara University of Science and Technology.

Exclusion Criteria:

* Exclude medical and nursing students in the pre-clinical years and those in non-clinical rotations at the time of the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Skills using the Scenario-execution-group test score | Immediately Post scenario execution
  This is a scenario specific score obtained from a multiple choice question (MCQ) test following execution of the scenario to measure. The MCQs are standard questions developed to accompany a given scenario. The maximum score is 100%. A scenario-execution-group test score of less than 60% will be a fail and a score of more than or equal to 60% will be a pass.

SECONDARY OUTCOMES:
Knowledge | Change in knowledge scores at 4 months from Baseline
  Knowledge will be measured using multiple choice questions (MCQs) and Investigators will use the Retrospective pre-post survey (RPP survey) to assess performance confidence among participants. In the RPP, the participant is asked to compare their performance after the intervention with that before the intervention. This assessment removes the bias of over or underestimating how much the participant knew before the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Santorini Data, MD, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Undecided
Data to be shared when necessary permissions have been obtained